CLINICAL TRIAL: NCT04208776
Title: Efficacy of Combination of Midodrine With Propranolol in Preventing First Bleed in Decompensated Cirrhotics With Severe Ascites: A Randomized Controlled Trial"
Brief Title: Efficacy of Combination of Midodrine With Propranolol in Preventing First Bleed in Decompensated Cirrhotics With Severe Ascites.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-27
Record Dates: First submitted 2019-12-12; First posted 2019-12-23 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Decompensated Cirrhosis; Severe Ascites
MeSH Terms: conditions — Ascites | interventions — Propranolol; Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midodrine+Propranolol (Experimental)
  Interventions: Drug: Propranolol; Drug: Midodrine
- Propranolol (Active Comparator)
  Interventions: Drug: Propranolol

INTERVENTIONS:
Drug: Propranolol — maximum tolerated dose of propranolol with initial dosage of 20mg once a day and uptitrating every 2nd day by 20 mg.
Drug: Midodrine — It will be started at 2.5mg TDS and will be uptitrated every 2nd day to a max of 10mg TDS to attain a MAP of atleast 70mm Hg and then uptitate the beta blocker simulataneously to attain the target heart rate
  Arms: Midodrine+Propranolol

SUMMARY:
Study population: Decompensated cirrhotics requiring primary prophylaxis with asciteswho are admitted to and attending the OPD at ILBS.

Study Design : A Randomized controlled trial Study period : August 2019 to December 2020 (1.5 Years) Intervention : Treatment naïve patients will be given Propranolol and dose will be titrated every 2ndday to attain a target heart rate of 55.

One group patients will be given maximum tolerated dose of propranolol with initial dosage of 20mg once a day and uptitrating every 2nd day by 20 mg.The patients who bleed will undergo EVL session.

To the other group Midodine will be added to Propranolol.It will be started at 2.5mg TDS and will be uptitrated every 2nd day to a max of 10mg TDS to attain a MAP of atleast 70mm Hg and then uptitate the beta blocker simulataneously to attain the target heart rate. The patients who bleed will undergo EVL session.

Monitoring and assessment :

The patient will be monitored every day. The patient will undergo physical examination, complete blood counts, at baseline, LFT, KFT, at every 2nd day and day 7 from the start of therapy.

Adverse effects : Bradycardia and hypotension due to beta blockers Stopping rule : Severe hyponatraemia (<125), low mean arterial pressure(<65) or cardiac output and increasing serum creatinine(>1.5) identifies more vulnerable patients among those with decompensated cirrhosis, in whom a dose reduction or temporal discontinuation of NSBB treatment will be considered.

ELIGIBILITY:
Inclusion Criteria:

Decompensated Child C cirrhotics with grade II-III requiring primary prophylaxis

Exclusion Criteria:

1. Spontaneous bacterial peritonitis
2. Hepatic Encephalopathy
3. Acute renal failure (S.Cr>1.5)
4. Hepatorenal syndrome
5. Hypertension
6. Coronary Artery Disease ; H/o arrhythmias, heart block
7. Urinary retention
8. Pheochromocytoma/thyrotoxicosis
9. Coronary Obstructive Pulmonary Disease
10. Hepatocellular Carcinoma
11. Pregnancy
12. Portal vein Thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-02-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Primary prevention of first variceal bleed in both groups | 1 year
  prevention of first variceal bleed is based on clinicallly

SECONDARY OUTCOMES:
Achievement of target heart rate (THR) of 55-60 or reduction by 25 % from baseline | Day 7
HVPG reduction in both groups | Day 90
  HVPG reduction by 20% from baseline
Survival in both groups | 1 year
Incidence of therapeutic paracentesis in both groups | Day 30
Incidence of therapeutic paracentesis in both groups | Day 90
Incidence of decrease in ascites by at least one grade in both groups | 3 months
Paracentesis induced circulatory dysfunction(PICD) in both groups | 1 year
  PICD is defined as Incidence of AKI and HE after paracentesis
Incidence of Hyponatremia in both groups | 1 year
  cut off for Hyponatremia is Sodium < 135
Episodes of bacterial infection in both groups | 1 year
  Bacterial infection will be identified by culture tests
Incidence of Hepatic Encephalopathy in both groups | 1 year
Incidence of Hepato Renal Syndrome in both groups | 1 year
Incidence of Acute Kidney Injury in both groups | 1 year
Incidence of Variceal bleed in both groups | 1 year
Number of TIPS (TransIntrahepatic Portosystemic Shunt) procedure done in both groups | 1 year
Number of patients who will receive diuretics in both groups | 1 year
Adverse effects of drugs in both groups | 1 year
Impact on portal, systemic and cardiac hemodynamics in both groups | 1 year
  For Portal and cardiac HVPG and right heart pressure studies will be done and for systemic blood pressure will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No